CLINICAL TRIAL: NCT02731989
Title: Comparison Between the Clinical Assessment of the Undescended Testis and Its' Ultrasonographic Size
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0090-16-MMC
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Undescended Testis
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study group: The surgeon will estimate the size difference between the undescended and the normally located testis. Independently the ultrasonographer will measure the true size of both testes in the study group.
- Control group: The same measurments will be done by the surgeon and the ultrasonographer on boys without cryptorchism.

SUMMARY:
In addition to the manual preoperative examination, the undescended testicle will be measured ultrasonographically. The compared data will help us to evaluate the routine need for preoperative ultrasonographic evaluation of the undescended testicle.

ELIGIBILITY:
Inclusion Criteria:

* Boys operated for unilateral cryptorchism

Exclusion Criteria:

* bilateral cryptorchism recurrent operation s/p inguinal operation

Ages: 1 Year to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Boys operated for unilateral cryptorchism
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-07-24 (Estimated); Primary Completion 2018-07-24 (Estimated); Study Completion 2019-07-24 (Estimated)

PRIMARY OUTCOMES:
The difference between the testicular size estimated by the surgeon and the actual ultrasonographic size | 3 years
  The difference between the testicular size estimated by the surgeon and the actual ultrasonographic size

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Centre, Kfar Saba, Israel